CLINICAL TRIAL: NCT05030623
Title: The Phosphodiesterase Inhibitor Tadalafil as an Adjunct to Antidepressants in Major Depressive Disorder Patients: Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Phosphodiesterase Inhibitor Tadalafil as an Adjunct to Antidepressants in Major Depressive Disorder Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15/2021NEUR
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil 5Mg Tab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 5Mg Tab — Tadalafil 5Mg Tab plus Fluoxetine 20 mg capsule
  Arms: Tadalafil
Drug: Placebo — Placebo Tab plus Fluoxetine 20 mg capsule
  Arms: Placebo

SUMMARY:
Antidepressant-like effects of tadalafil to its ability to modulate transduction pathways responsible for neuroplasticity. Treatment with tadalafil was shown to be PKG-dependent and lead to increased expression of cGMP, pCREB, BDNF and VGF in the hippocampus and prefrontal cortex (PFC), brain areas relevant to mood disorders pathophysiology. Low-dose tadalafil improved both depressive symptoms in patients with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 18 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).

Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

Patients with bipolar I or bipolar II disorder Patients with personality disorders Patients with eating disorders Patients with substance dependence or abuse Patients with concurrent active medical condition Patients with history of seizures Patients with history of receiving Electroconvulsive therapy (ECT) Patients with inflammatory disorders Patients with allergy or contraindications to the used medications Patients with finally pregnant or lactating females Cardiovascular disorders Severe renal impairment: creatinine clearance of ≤ 25 ml/min Moderate or severe hepatic impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 12 weeks
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
Effect on biological markers | At baseline and after 12 weeks of intervention
  Serum level of tumor necrosis factor alpha (TNF-α), Interleukin-6 (IL-6), and brain derived neurotrophic factor (BDNF) were measured at the baseline and after the treatment to evaluate the biological effects of the used medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF